CLINICAL TRIAL: NCT04220515
Title: Phase IV Safety Monitoring Study of Inactivated Poliomyelitis Vaccine Made From Sabin Strain
Brief Title: Inactivated Poliomyelitis Vaccine Made From Sabin Strain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Shanghai Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20170416
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inactivated Poliomyelitis Vaccine Made From Sabin Strain (Experimental): Primary 3-dose of sIPV and booster 1 dose of sIPV
  Interventions: Biological: Inactivated Poliomyelitis Vaccine Made From Sabin Strain

INTERVENTIONS:
Biological: Inactivated Poliomyelitis Vaccine Made From Sabin Strain — Type I D antigen 30DU;Type II D antigen 32DU;Type III D antigen 45 DU

SUMMARY:
This study includes both active and passive safety monitoring in large pupulations for the phase IV safety monitoring study of Inactivated Poliomyelitis Vaccine Made From Sabin Strain (sIPV).

DETAILED DESCRIPTION:
For active safety monitoring in expanding populations, a total of 20,019 participants in Shanghai CDC have been enrolled in accordance with GCP for close safety monitoring for immediate adverse events and telephone or visiting follow-up (30 min, 24h, 3d, 7d, 14d, 30d) For passive safety monitoring in larger populations, the purpose is to observe rare adverse events after primary and booster immunization with sIPV by passive safety surveillance via AEFI monitoring system in Shanghai CDC. A total of 29,712 infants have been enrolled, and the adverse events of the participates have been collected via AEFI monitoring system and evaluated after 3-dose sIPV for primary immunization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants of 2 months of age
* The legal identity certificate (birth/household register) and vaccination certificate of the participants can be provided, and the legal guardian can provide the legal identity certificate (identity card).
* Guardians are able to understand the experimental vaccine, volunteer to participate in the study and sign informed consent for participation.
* Guardians are capable of using thermometer, graduated scale, filling diary card and contact card.
* Participants are not vaccinated with polio vaccine and immunoglobulin (except for Hepatitis b specific immunoglobulin) after birth, no vaccination of live vaccine within 28 days before enrollment and no vaccination of inactivated vaccine within 14 days before enrollment.
* Participants or guardians are able to obey and follow all study instructions, complete all the monitoring, and cooperate to complete collection of blood sample.
* Axillary temperature ≤37℃

Exclusion Criteria:

* Allergic to any active substance, inactive substance or materials used during production such as kanamycin.
* Patients with fever or acute disease.
* Have thrombocytopenia or hemorrhagic diseases
* Patients undergoing immunosuppressive therapy or immunodeficiency
* Have uncontrolled epilepsy or other progressive neurological disorders
* Other situations that the investigator consider as non-eligible

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49731 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Safety monitoring | 30 days post inoculation
  Active and passive monitoring for local and systemic adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, Principal Investigator — Disease prevention and control center of Shanghai
Locations (1):
- Disease prevention and control center of Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Participants do not agree to share the individual data.

REFERENCES:
- [Derived] Jiang R, Liu X, Sun X, Wang J, Huang Z, Li C, Li Z, Zhou J, Pu Y, Ying Z, Yin Q, Zhao Z, Zhang L, Lei J, Bao W, Jiang Y, Dou Y, Li J, Yang H, Cai W, Deng Y, Che Y, Shi L, Sun M. Immunogenicity and safety of the inactivated poliomyelitis vaccine made from Sabin strains in a phase IV clinical trial for the vaccination of a large population. Vaccine. 2021 Mar 1;39(9):1463-1471. doi: 10.1016/j.vaccine.2021.01.027. Epub 2021 Jan 22. PMID 33487470